CLINICAL TRIAL: NCT06328075
Title: Artificial Intelligence to Assist the Echocardiographic Identification of Transthyretin Cardiac Amyloidosis
Acronym: AI-ATTR-ECHO
Status: Recruiting | Type: Observational
Sponsor: Algalarrondo Vincent (Other)
Collaborators: Bichat Hospital (Other); Bioquantis (Unknown)
Responsible Party: Sponsor-Investigator, Algalarrondo Vincent, Principal Investigator, Director of the referral center CRMR -CERAMIC CARDIO, Bichat Hospital
Organization: Bichat Hospital (Other)
Other Study IDs: AI-ATTR-ECHO; 20211029191554 (Other: registre général des traitements de l'APHP)
Record Dates: First submitted 2024-03-12; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Amyloid Cardiomyopathy; Transthyretin Amyloid Cardiomyopathy; Transthyretin Cardiac Amyloidosis
Keywords: echocardiography; artificial intelligence; Transthyretin Amyloid Cardiomyopathy
MeSH Terms: conditions — Amyloid Neuropathies, Familial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transthyretin cardiac amyloidosis (ATTR-CM): Patients with an ATTR-CM and undergoing a transthoracic echocardiography
  Interventions: Other: non interventional study
- Controls: Patients without cardiac amyloidosis undergoing transthoracic echocardiography as part of cardiological follow-up
  Interventions: Other: non interventional study

INTERVENTIONS:
Other: non interventional study — non interventional study

SUMMARY:
The goal of this study is to develop an algorithm using artificial intelligence (AI) to assist identification of potential ATTR-CM cases using routine transthoracic echocardiography.

The main questions it aims to answer are:

* is the algorithm able to diagnose ATTR-CM
* is the algorithm able to diagnose different types of ATTR-CM (ATTRv, ATTRwt)

This is a non interventional study. Participant' echocardiographies will be, after deidentification, used to train, valid and test the algorithm.

DETAILED DESCRIPTION:
Transthyretin (TTR) amyloidosis is a serious systemic disease affecting multiple target organs including the peripheral nervous system, heart, and kidney. In the absence of treatment, the median survival for symptomatic forms with cardiac involvement is 3 to 4 years.

In recent years, new treatments have proven their effectiveness in transthyretin amyloidosis, making it possible to slow the progression of neuropathy and cardiac damage. These treatments seem particularly effective when they are initiated at an early stage of the disease.

It is therefore necessary to establish the diagnosis as early as possible in order to benefit the most from the treatment. However, during the clinical examination, the electrocardiogram or the routine echocardiography, the signs evoking cardiac amyloidosis are not specific. The initial diagnosis is therefore often difficult, missed or delayed and the median time between the first symptoms and the initiation of treatment is approximately 3 years.

It is therefore the initial phase of diagnosis that must be improved in a sufficiently sensitive and specific manner to detect potential cases early while avoiding unnecessary examinations in the event of a low probability.

The objective of the study is to develop and validate a tool to assist the screening of cardiac transthyretin amyloidosis, from standard echocardiography, without the need for active participation of the cardiologist in the diagnostic process. This diagnostic contribution will allow the cardiologist to evoke the diagnosis of cardiac amyloidosis and to consider additional explorations.

ELIGIBILITY:
ATTR-CM patients:

Inclusion Criteria:

* Cardiac transthyretin amyloidosis diagnosed on the classic criteria:

  1. Absence of monoclonal immunoglobulin AND
  2. Presence of a bisphosphonate scintigraphy with enhancement in the cardiac area OR

  2-Presence of a cardiac biopsy showing transthyretin (Congo red positive) cardiac amyloidosis (demonstrated either by immunostaining or by mass spectrometry) OR 3-Presence of a peripheral biopsy showing transthyretin amyloidosis (see above) associated with cardiac infiltration (parietal thickness >12mm without other cause of cardiac hypertrophy)
* No opposition to research

Non-inclusion criteria:

* Another cause of cardiac amyloidosis: AL AA amyloidosis…
* Mixed heart disease with associated presence of non-amyloid heart disease (ischemic heart disease, dilated, etc.)

Control patients:

Inclusion criteria:

* Indication for transthoracic echocardiography as part of cardiological follow-up
* Patient affiliated with social security
* Patient's agreement to participate in the research and signature of the consent form.
* Technical conditions of the examination and echogenicity allowing acquisition of good quality echocardiographic images, allowing post processing

Non-inclusion criteria:

* Presence of cardiac amyloidosis as defined above
* Presence of transthyretin amyloidosis even without demonstrated cardiac involvement
* Patient monitored for asymptomatic transthyretin mutation
* Minor patient or patient unable to give their consent (unconscious patient, under guardianship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The ATTR-CM cohort will be recruited in referral tertiary centers for cardiac amyloidosis The Control cohort will be recruited in the same centers from patients presenting an indication for transthoracic echocardiography as part of cardiological follow-up
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Building and validating the diagnostic performance metrics curves of the AI algorithm to diagnose ATTR-CM : | year 1
  To develop and validate a tool using artificial intelligence an algorithm that will improve the automatic detection on routinely acquired echocardiography images of aspects suggestive of transthyretin amyloidosis.
  A confusion matrix will be built and the following diagnostic performance metrics be computed:
  * receiver operating characteristic curve (ROC) and area under curve (AUC) of the ROC : AUROC
  * Precision recall curve (PR) and area under curve (AUC) of the PR curve : AUC-PR
Building and validating the diagnostic performance metrics of the AI algorithm to diagnose ATTR-CM : | year 1
  To develop and validate a tool using artificial intelligence an algorithm that will improve the automatic detection on routinely acquired echocardiography images of aspects suggestive of transthyretin amyloidosis ATTR.
  A confusion matrix will be built and the following diagnostic performance metrics be computed:
  Accuracy, Sensitivity or Recall, Specificity, False positive rate, False Negative Rate, Precision (all are expressed as ratio)

SECONDARY OUTCOMES:
Building and validating the diagnostic performance metrics of the AI algorithm to diagnose ATTRwt-CM : | year 1
  To develop and validate a tool using artificial intelligence an algorithm that will improve the automatic detection on routinely acquired echocardiography images of aspects suggestive of transthyretin amyloidosis.
  A confusion matrix will be built and the following diagnostic performance metrics be computed:
  Accuracy, Sensitivity or Recall, Specificity, False positive rate, False Negative Rate, Precision (all are expressed as ratio)
Building and validating the diagnostic performance metrics of the AI algorithm to diagnose ATTRv-V122I-CM : | year 1
  To develop and validate a tool using artificial intelligence an algorithm that will improve the automatic detection on routinely acquired echocardiography images of aspects suggestive of transthyretin amyloidosis.
  A confusion matrix will be built and the following diagnostic performance metrics be computed:
  Accuracy, Sensitivity or Recall, Specificity, False positive rate, False Negative Rate, Precision (all are expressed as ratio)
Building and validating the diagnostic performance metrics of the AI algorithm to diagnose ATTRv-CM : | year 1
  To develop and validate a tool using artificial intelligence an algorithm that will improve the automatic detection on routinely acquired echocardiography images of aspects suggestive of transthyretin amyloidosis.
  A confusion matrix will be built and the following diagnostic performance metrics be computed:
  Accuracy, Sensitivity or Recall, Specificity, False positive rate, False Negative Rate, Precision (all are expressed as ratio)
Building and validating the diagnostic performance metrics of the AI algorithm to differentiate ATTR-CM from LV hypertrophy (LVH) : | year 1
  To develop and validate a tool using artificial intelligence an algorithm that will improve the automatic detection on routinely acquired echocardiography images of aspects suggestive of transthyretin amyloidosis from LVH.
  A confusion matrix will be built and the following diagnostic performance metrics be computed:
  Accuracy, Sensitivity or Recall, Specificity, False positive rate, False Negative Rate, Precision (all are expressed as ratio)
Building and validating the diagnostic performance metrics curves of the AI algorithm to diagnose ATTRwt-CM : | year 1
  To develop and validate a tool using artificial intelligence an algorithm that will improve the automatic detection on routinely acquired echocardiography images of aspects suggestive of transthyretin amyloidosis (ATTRwt subgroup).
  A confusion matrix will be built and the following diagnostic performance metrics be computed:
  * receiver operating characteristic curve (ROC) and area under curve (AUC) of the ROC : AUROC
  * Precision recall curve (PR) and area under curve (AUC) of the PR curve : AUC-PR
Building and validating the diagnostic performance metrics curves of the AI algorithm to diagnose ATTRv-V122I-CM : | year 1
  To develop and validate a tool using artificial intelligence an algorithm that will improve the automatic detection on routinely acquired echocardiography images of aspects suggestive of transthyretin amyloidosis (ATTRv-V122I subgroup).
  A confusion matrix will be built and the following diagnostic performance metrics be computed:
  * receiver operating characteristic curve (ROC) and area under curve (AUC) of the ROC : AUROC
  * Precision recall curve (PR) and area under curve (AUC) of the PR curve : AUC-PR
Building and validating the diagnostic performance metrics curves of the AI algorithm to diagnose ATTRv-CM : | year 1
  To develop and validate a tool using artificial intelligence an algorithm that will improve the automatic detection on routinely acquired echocardiography images of aspects suggestive of transthyretin amyloidosis (ATTRv-subgroup).
  A confusion matrix will be built and the following diagnostic performance metrics be computed:
  * receiver operating characteristic curve (ROC) and area under curve (AUC) of the ROC : AUROC
  * Precision recall curve (PR) and area under curve (AUC) of the PR curve : AUC-PR
Building and validating the diagnostic performance metrics curves of the AI algorithm to differentiate ATTR-CM from LV hypertrophy (LVH) : | year 1
  To develop and validate a tool using artificial intelligence an algorithm that will improve the automatic detection on routinely acquired echocardiography images of aspects suggestive of transthyretin amyloidosis (ATTRv-subgroup) in a subset of patients with LVH.
  A confusion matrix will be built and the following diagnostic performance metrics be computed:
  * receiver operating characteristic curve (ROC) and area under curve (AUC) of the ROC : AUROC
  * Precision recall curve (PR) and area under curve (AUC) of the PR curve : AUC-PR

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Steg, MD, PhD, Study Chair — Bichat Hospital
Locations (1):
- Bichat, Paris, France

IPD SHARING:
Plan to Share IPD: No
Investigators will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon reasonable request from qualified researchers, and subject to certain criteria, conditions, and exceptions.